CLINICAL TRIAL: NCT07294495
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Effect of Henagliflozin on Myocardial Fibrosis Burden in Patients With Non-Obstructive Hypertrophic Cardiomyopathy Using 68Ga/18F-FAPI PET/CMR
Brief Title: Effect of Henagliflozin on Myocardial Fibrosis in Non-Obstructive HCM: A Randomized, Double-Blind, Placebo-Controlled Trial Using 68Ga/18F-FAPI PET/CMR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025286
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: HCM - Hypertrophic Cardiomyopathy
Keywords: PET/MR; FAPI; Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — henagliflozin; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Intervention Model Description: This study employs a two-arm, parallel-group, randomized controlled trial model. Eligible participants are randomly assigned in a 1:1 ratio to one of two parallel treatment arms. Both arms receive their assigned intervention (active drug or matched placebo) concurrently over the same fixed period of 6 months, followed by a common follow-up schedule. The outcomes are compared between these independent, parallel groups at pre-defined time points.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind trial where the participant, the care provider (investigator), and the outcomes assessor (including imaging analysts and statisticians) are all masked to group assignment. The active drug (Henagliflozin) and the matched placebo are identical in appearance, packaging, and labeling. The randomization code is maintained by an independent central pharmacy and the Interactive Web Response System. Unblinding occurs only in medical emergencies or after database lock.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Henagliflozin (SGLT2 Inhibitor) (Experimental): Participants randomized to this arm will receive a once-daily oral dose of Henagliflozin (10 mg tablet) for a total intervention period of 6 months. Henagliflozin is a selective sodium-glucose cotransporter 2 (SGLT2) inhibitor. All participants will continue their stable standard background therapy for hypertrophic cardiomyopathy throughout the study.
  Interventions: Drug: Henagliflozin (SGLT2 Inhibitor)
- Placebo (Placebo Comparator): Participants randomized to this arm will receive a once-daily oral dose of a matching placebo tablet for a total intervention period of 6 months. The placebo is identical in appearance, packaging, and administration schedule to the active drug. All participants will continue their stable standard background therapy for hypertrophic cardiomyopathy throughout the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Henagliflozin (SGLT2 Inhibitor) — This intervention involves the oral administration of Henagliflozin, a selective sodium-glucose cotransporter 2 (SGLT2) inhibitor, at a dose of 10 mg once daily for a period of 6 months. Henagliflozin is provided as a film-coated tablet identical in appearance to the matched placebo used in the control arm. The intervention is administered in a double-blind manner as an add-on to stable standard background therapy for non-obstructive hypertrophic cardiomyopathy. This study specifically investigates the potential anti-fibrotic effects of Henagliflozin on active myocardial fibrosis, as quantified by novel FAPI PET/CMR imaging, in a patient population without diabetes mellitus.
  Arms: Henagliflozin (SGLT2 Inhibitor)
Drug: Placebo — This intervention involves the oral administration of a matched placebo tablet once daily for a period of 6 months. The placebo is manufactured to be identical in appearance (size, shape, color, coating), packaging, and administration schedule to the active comparator, Henagliflozin 10 mg tablet. It contains no active pharmaceutical ingredient. The intervention is administered in a double-blind manner as an add-on to stable standard background therapy for non-obstructive hypertrophic cardiomyopathy, serving as the control to isolate and evaluate the specific pharmacological effects of the SGLT2 inhibitor.
  Arms: Placebo

SUMMARY:
his is a single-center, randomized, double-blind, placebo-controlled clinical trial designed to evaluate the effect of Henagliflozin (an SGLT2 inhibitor) on myocardial fibrosis burden in patients with non-obstructive hypertrophic cardiomyopathy (nHCM). The study will use 68 68 Ga/ 18 18 F-FAPI PET/CMR imaging to quantitatively assess changes in active fibroblast activity after 6 months of treatment. A total of 150 eligible adult patients with nHCM (FAPI-positive at baseline, NYHA class I-III) will be enrolled and randomized in a 1:1 ratio to either the Henagliflozin group (10 mg once daily) or the placebo group for a 6-month treatment period. The primary endpoint is the change in myocardial FAPI target-to-background ratio (ΔTBR) at 6 months. Secondary endpoints include changes in FAPI SUVmax, FAPI burden percentage (FAV%), cardiac structure and function parameters, 6-minute walk distance, NYHA classification, NT-proBNP levels, and quality-of-life scores. Exploratory analyses will assess clinical events over 12 months, such as heart failure hospitalization, atrial fibrillation, ventricular arrhythmias, and cardiovascular death. The study employs stratified block randomization based on baseline FAPI burden, central randomization and blinding via IWRS, independent core laboratory imaging evaluation, and an intention-to-treat analytical approach. It aims to provide early evidence for the anti-fibrotic effect of Henagliflozin in nHCM and to validate FAPI-PET/CMR as an imaging biomarker for fibrosis activity.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, placebo-controlled clinical trial designed to evaluate the effect of Henagliflozin, an SGLT2 inhibitor, on myocardial fibrosis burden in patients with non-obstructive hypertrophic cardiomyopathy. The study will utilize integrated Gallium-68 or Fluorine-18 labeled FAPI PET/CMR imaging to quantitatively assess changes in active fibroblast activity following six months of treatment. A total of 150 eligible adult patients with non-obstructive hypertrophic cardiomyopathy, who are FAPI-positive at baseline and classified as NYHA functional class I to III, will be enrolled. Participants will be randomized in a one-to-one ratio to receive either Henagliflozin 10 mg once daily or a matching placebo for a treatment period of six months.

The primary endpoint of the study is the change in myocardial FAPI target-to-background ratio from baseline to six months. Secondary endpoints include changes in other FAPI parameters such as SUVmax and FAPI-active volume percentage, as well as changes in cardiac structure and function parameters assessed by CMR, six-minute walk distance, NYHA functional class, NT-proBNP levels, and quality of life scores. Furthermore, exploratory analyses will assess clinical events over a 12-month period, including heart failure hospitalization, atrial fibrillation, ventricular arrhythmias, and cardiovascular death.

The trial employs a stratified block randomization method based on baseline FAPI burden, with central randomization and blinding maintained through an interactive web response system. All imaging data will be evaluated by an independent core laboratory to ensure objectivity, and statistical analyses will adhere to the intention-to-treat principle. This study aims to generate early evidence regarding the potential anti-fibrotic effect of Henagliflozin in non-obstructive hypertrophic cardiomyopathy and to validate FAPI-PET/CMR as a promising imaging biomarker for monitoring myocardial fibrosis activity.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older, regardless of gender.
2. Meets the diagnostic criteria for non-obstructive hypertrophic cardiomyopathy (HCM):

   * Confirmed diagnosis of HCM by cardiac magnetic resonance (CMR) or echocardiography (left ventricular wall thickness ≥15 mm, or ≥13 mm in the presence of a family history of HCM).
   * Exclusion of patients in whom left ventricular hypertrophy is primarily attributable to hypertensive heart disease, as assessed by a cardiology specialist based on clinical and imaging evidence.
   * Exclusion of other identifiable causes of secondary myocardial hypertrophy (e.g., valvular heart disease, storage cardiomyopathies).
   * Left ventricular outflow tract (LVOT) gradient <30 mmHg at rest or under provocation, as assessed by echocardiography or CMR.
3. Willing to undergo FAPI PET/CMR examination and complete imaging evaluations.
4. Baseline FAPI PET/CMR scan shows positive FAPI uptake: myocardial FAPI target-to-background ratio (TBR) ≥1.3, using the ascending aorta blood pool as the background reference.
5. Capable of understanding and signing the informed consent form, and agrees to participate in the study, accept randomization, and comply with follow-up visits.
6. New York Heart Association (NYHA) functional class I-III.

Exclusion Criteria:

1. Significant left ventricular outflow tract obstruction (resting or provoked LVOT pressure gradient ≥30 mmHg).
2. Coexistence of other identifiable causes of myocardial hypertrophy, including:

   * Predominant or persistent hypertensive heart disease;
   * Severe aortic stenosis or other significant valvular heart disease;
   * Infiltrative or storage cardiomyopathies (e.g., Fabry disease, amyloidosis);
   * Ischemic heart disease (e.g., severe coronary artery disease).
3. Overt decompensated heart failure or NYHA functional class IV.
4. Unstable, serious arrhythmias (e.g., sustained ventricular tachycardia, recent cardioversion for atrial fibrillation).
5. Recent (within 3 months) cardiac surgery or interventional procedure.
6. ALT or AST >3 times the upper limit of normal (ULN), OR total bilirubin (Tbil) >2 times ULN, OR ketonuria/ketonemia, OR eGFR <30 mL/min/1.73m², OR creatine kinase (CK) >3 times ULN.
7. Concurrent other severe systemic disease with a life expectancy of less than 1 year.
8. Pregnant or breastfeeding women.
9. History of allergy to the study drug or any contraindication to its use.
10. Any other condition deemed by the investigator to make the subject unsuitable for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-07 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Myocardial FAPI Target-to-Background Ratio (ΔTBR) | From baseline to 6 months post-intervention
  The primary outcome is the change in myocardial FAPI uptake quantified by the target-to-background ratio (TBR) on FAPI PET/CMR imaging. TBR is calculated as the ratio of the mean standardized uptake value (SUVmean) in the myocardium to that in the ascending aortic blood pool. The difference in TBR from baseline to 6 months post-intervention (ΔTBR) will be compared between the Henagliflozin and placebo groups. This measure directly reflects changes in active fibroblast activity and myocardial fibrosis burden.

SECONDARY OUTCOMES:
Change in Myocardial FAPI Maximum Standardized Uptake Value (ΔSUVmax) | From baseline to 6 months post-intervention
  This outcome measures the change in the maximum standardized uptake value of FAPI within the myocardium, reflecting the activity of the most intense focal fibrotic lesion. It is quantified from the same FAPI PET/CMR images used for the primary outcome.
Change in FAPI Activity Volume Percentage (ΔFAV%) | From baseline to 6 months post-intervention
  This outcome measures the percentage change in myocardial volume exhibiting active fibrosis. It is calculated by applying a standardized SUV threshold (e.g., SUV ≥ 1.3) to the FAPI PET images to define FAPI-positive voxels and expressing their volume as a percentage of the total left ventricular myocardium volume.
Change in Left Ventricular Ejection Fraction (ΔLVEF) | From baseline to 6 months post-intervention
  This outcome assesses the change in global left ventricular systolic function, measured as the percentage of blood ejected from the left ventricle with each contraction, using cardiac magnetic resonance imaging.
Change in Left Ventricular Mass Index (ΔLVMi) | From baseline to 6 months post-intervention
  This outcome measures the change in left ventricular myocardial mass, adjusted for body surface area, as an indicator of regression or progression of myocardial hypertrophy, assessed via cardiac magnetic resonance.
Change in Late Gadolinium Enhancement Extent (ΔLGE) | From baseline to 6 months post-intervention
  This outcome quantifies the change in the volume or mass of replacement (scar) fibrosis within the left ventricle using the late gadolinium enhancement technique on cardiac magnetic resonance.
Change in Global Longitudinal Strain (ΔGLS) | From baseline to 6 months post-intervention
  This outcome measures the change in myocardial deformation during contraction, specifically the peak systolic longitudinal strain averaged across all left ventricular segments, assessed by CMR feature-tracking. It is a sensitive marker of early myocardial dysfunction.
Change in 6-Minute Walk Distance (Δ6MWD) | From baseline to 6 months post-intervention
  This outcome measures the change in functional exercise capacity by recording the total distance (in meters) a participant can walk on a flat, hard surface in 6 minutes, following standardized guidelines.
Change in New York Heart Association (NYHA) Functional Class | From baseline to 6 months post-intervention
  This outcome measures the proportion of participants with an improvement (e.g., reduction by one or more classes) in their NYHA functional class, which categorizes the severity of heart failure symptoms and physical limitations.
Change in Serum NT-proBNP Level | From baseline to 6 months post-intervention
  This outcome measures the absolute or percent change in serum N-terminal pro-B-type natriuretic peptide concentration, a biomarker associated with cardiac wall stress and heart failure severity.
Change in Quality of Life Total Score (SF-36) | From baseline to 6 months post-intervention
  This outcome measures the change in overall health-related quality of life using the total score of the 36-Item Short Form Health Survey (SF-36), which covers physical and mental health domains.

OTHER OUTCOMES:
Significant Worsening of Cardiac Function or Onset of Heart Failure | Throughout the 12-month study period
  This outcome is a composite endpoint capturing clinically meaningful deterioration in heart failure status, defined as any of the following: worsening of NYHA functional class by one or more grades, hospitalization primarily due to heart failure, or a decline in 6-minute walk distance of ≥30 meters from baseline.
New Onset or Recurrence of Atrial Fibrillation/Atrial Flutter | Throughout the 12-month study period
  This outcome records the occurrence of newly diagnosed or recurrent episodes of atrial fibrillation or atrial flutter, confirmed by standard 12-lead electrocardiogram, Holter monitoring, or other clinically documented evidence during follow-up.
Sustained or Non-Sustained Ventricular Tachycardia | Throughout the 12-month study period
  This outcome captures episodes of ventricular tachycardia, defined as sustained (lasting ≥30 seconds or requiring termination due to hemodynamic compromise) or non-sustained (≥3 consecutive ventricular beats at a rate >100 bpm, lasting <30 seconds), documented by ECG or cardiac monitoring.
Sudden Cardiac Death or Cardiac Arrest | Throughout the 12-month study period
  This outcome records fatal events adjudicated as sudden cardiac death (unexpected death within 1 hour of symptom onset in a stable patient, or unwitnessed death without other explanation) or non-fatal cardiac arrest requiring resuscitation.
Cardiac-Related Hospitalization | Throughout the 12-month study period
  This outcome measures hospital admissions primarily due to a cardiovascular cause, including but not limited to worsening heart failure, arrhythmia, acute coronary syndrome, or other cardiac complications, as determined by clinical adjudication.
Cardiovascular Death | Throughout the 12-month study period
  This outcome captures death attributable to cardiovascular causes, including fatal myocardial infarction, heart failure, stroke, arrhythmia, or other direct cardiac etiologies, as adjudicated by an independent clinical endpoint committee.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) collected and generated in this study, including de-identified datasets, will not be made publicly available. The data are primarily used to fulfill the pre-specified objectives of this investigator-initiated trial. Data may be disclosed to regulatory authorities upon request for audit or review purposes, or for validating key findings in future scientific collaborations under strict data use agreements. However, there is no current plan for systematic public sharing or deposition in a public repository.